CLINICAL TRIAL: NCT00363584
Title: A Randomised Clinical Trial Evaluating Adjuvant Chemotherapy With Capecitabine Compared to Expectant Treatment Alone (Observation) Following Surgery for Biliary Tract Cancer
Brief Title: Capecitabine or Observation After Surgery in Treating Patients With Biliary Tract Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000492266; CRUK-HE3002; EU-20629; EUDRACT-2005-003318-13; ISRCTN72785446; CRUK-BILCAP; CRUK-BIBF1120
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2011-10

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Liver Cancer
Keywords: localized resectable adult primary liver cancer; cholangiocarcinoma of the extrahepatic bile duct; cholangiocarcinoma of the gallbladder; adenocarcinoma of the gallbladder; adenocarcinoma with squamous metaplasia of the gallbladder; anaplastic carcinoma of the gallbladder; localized gallbladder cancer; localized extrahepatic bile duct cancer; squamous cell carcinoma of the gallbladder; adult primary cholangiocellular carcinoma
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Liver Neoplasms | interventions — Capecitabine; Watchful Waiting; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: capecitabine
Other: clinical observation
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving capecitabine after surgery may kill any tumor cells that remain after surgery. Sometimes, after surgery, the tumor may not need more treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether capecitabine is more effective than observation in treating biliary tract cancer.

PURPOSE: This randomized phase III trial is studying capecitabine to see how well it works compared with observation in treating patients with biliary tract cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether adjuvant chemotherapy with capecitabine has any effect on 2-year survival compared to expectant treatment alone (observation) in patients who have undergone a macroscopically complete surgical resection of a biliary tract cancer.

Secondary

* To compare capecitabine versus observation in terms of 5-year survival, relapse-free survival, toxicity, quality of life, and health economics.

OUTLINE: This is a multicenter, prospective, randomized study. Patients are stratified according to surgical center, disease site (hilar/extrahepatic cholangiocarcinoma vs intrahepatic cholangiocarcinoma vs gallbladder vs intrapancreatic/common bile duct), type of resection (R0 vs R1), and ECOG performance status (0 vs 1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral capecitabine twice a day on days 1-14. Treatment repeats every 3 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo expectant treatment (observation). Quality of life is assessed at baseline, every 3 months for 1 year, and then every 6 months for 1 year.

All patients are followed for up to 5 years post-randomization.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 360 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed biliary tract cancer (including intrahepatic or extrahepatic/hilar cholangiocarcinoma or muscle invasive gallbladder cancer or cancer of the distal bile duct)

  * Must have undergone a radical surgical approach which includes liver resection, pancreatic resection, or less commonly both
  * Patients with pathological evidence of microscopic involvement of the margins of the excised specimen are eligible as long as resection is macroscopically complete
* Must be able to start treatment within 12 weeks of surgery
* No pancreatic or periampullary cancer
* No mucosal gallbladder cancer

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Urea < 1.5 times upper limit of normal (ULN)
* Creatinine < 1.5 times ULN
* Glomerular filtration rate ≥ 60 mL/min (if < 60 mL/min, adequate renal function for capecitabine must be confirmed by isotope EDTA)
* Hemoglobin ≥ 10 g/dL
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 3 times ULN
* ALT and AST ≤ 5 times ULN
* Adequate surgical biliary drainage with no evidence of infection
* Not pregnant or nursing
* Negative pregnancy test for women of childbearing age and childbearing potential
* Fertile patients must use effective contraception during study treatment and for at least 3 months after study treatment has ended
* Must provide written informed consent
* No history of other malignant diseases within the past 5 years other than adequately treated nonmelanoma skin cancer or in situ carcinoma of the uterine cervix
* No serious co-existing medical condition likely to interfere with protocol treatment, including a potential serious infection
* No evidence of significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial
* No psychological, familial, sociological, or geographical factors considered likely to preclude study compliance
* No other serious uncontrolled medical conditions
* No unresolved biliary tree obstruction

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Completely recovered from prior surgery
* No use of other investigational agents within 28 days prior to and during study treatment
* No prior chemotherapy or radiotherapy for biliary tract cancer
* No other concurrent anticancer chemotherapy, radiotherapy, or investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2006-03; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Survival at 2 years

SECONDARY OUTCOMES:
Survival at 5 years
Relapse-free survival
Toxicity
Quality of life
Health economics

CONTACTS AND LOCATIONS:
Overall Officials: Clive Stubbs — Cancer Research Campaign Clinical Trials Centre
Locations (46):
- United Kingdom (46):
  - Basildon University Hospital, Basildon, England
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Cancer Research UK Clinical Trials Unit - Birmingham, Birmingham, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Walsgrave Hospital, Coventry, England
  - Princess Alexandra Hospital, Essex, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Calderdale Royal Hospital, Halifax, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Cancer Research UK Clinical Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Leicester General Hospital, Leicester, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Aintree University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Helen Rollason Cancer Care Centre at North Middlesex Hospital, London, England
  - UCL Cancer Institute, London, England
  - St. Thomas' Hospital, London, England
  - King's College Hospital, London, England
  - Royal Marsden - London, London, England
  - Hammersmith Hospital, London, England
  - University College of London Hospitals, London, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital, Manchester, England
  - North Manchester General Hospital - Penine Actute Hospitals Trust, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Freeman Hospital, Newcastle upon Tyne, England
  - St. Mary's Hospital, Newport, England
  - Nottingham City Hospital, Nottingham, England
  - Derriford Hospital, Plymouth, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth Hants, England
  - Alexandra Healthcare NHS, Redditch, Worcestershire, England
  - Salisbury District Hospital, Salisbury, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Yeovil District Hospital, Yeovil, England
  - Ninewells Hospital, Dundee, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Perth Royal Infirmary, Perth, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales

REFERENCES:
- [Derived] Keller HR, Fluke L, Forrester JA, Wolf RF. Identifying Indications for Neoadjuvant Therapy in Cholangiocarcinoma. Oncology (Williston Park). 2024 Apr 11;38(4):160-162. doi: 10.46883/2024.25921017. PMID 38661512